CLINICAL TRIAL: NCT06644378
Title: A Phase 1, Open-label, 2-part Study of the Absorption, Metabolism, and Excretion, and Absolute Bioavailability of [14C]-LY3866288 in Healthy Participants
Brief Title: A Study of [14C]-LY3866288 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18885; J4G-OX-JZVB (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Radioactive; ADME; Disposition; Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: [14C]-LY3866288 (Experimental): Single dose of [¹⁴C]-LY3866288 administered orally.
  Interventions: Drug: [14C]-LY3866288
- Part B: LY3866288 + [14C]-LY3866288 (Experimental): Single dose of LY3866288 administered orally followed by a single dose of [¹⁴C]-LY3866288 administered intravenously (IV).
  Interventions: Drug: LY3866288; Drug: [14C]-LY3866288

INTERVENTIONS:
Drug: [14C]-LY3866288 — Administered orally.
  Arms: Part A: [14C]-LY3866288
Drug: LY3866288 — Administered orally.
  Arms: Part B: LY3866288 + [14C]-LY3866288
Drug: [14C]-LY3866288 — Administered IV.
  Arms: Part B: LY3866288 + [14C]-LY3866288

SUMMARY:
The main purpose of this study is to evaluate how much of the study drug (LY3866288), administered as a single dose that has the radioactive substance 14C incorporated into it, passes from blood into urine, feces and expired air in healthy participants. The study will also measure how much of the study drug gets into the bloodstream when taken orally, compared to when injected directly into the vein, how its broken down, and how long it takes the body to get rid of it. The study will also evaluate the safety and tolerability of LY3866288.The study is conducted in two parts. The study is expected to last approximately 68 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy determined by medical history, physical examination, 12-lead ECGs, vital signs measurements, and clinical laboratory evaluations at screening and/or check-in by the investigator
* Have Body mass index between 18.0 and 32.0 kg/m^2 (kilograms per meter squared)
* Male participants who are infertile via bilateral orchiectomy or vasectomy
* Female participants (non-childbearing potential only for Part A) who follow standard contraceptive methods

Exclusion Criteria:

* Female participants who are lactating or pregnant
* Have history of alcohol and/or drug abuse within 2 years prior to screening
* Have history or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Have history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Part A, Fraction of [14C]-LY3866288 Dose Excreted in Urine (Feur) Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 21 postdose
Part A, Fraction of Dose [14C]-LY3866288 Excreted in Feces Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 21 postdose
Part B, Absolute Bioavailability (Fabs) of LY3866288 | Predose up to Day 9 postdose

SECONDARY OUTCOMES:
Part A: Pharmacokinetics (PK): Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of LY3866288 in Plasma Following a Single Oral Dose of [14C]-LY3866288 | Predose up to Day 7 postdose
Part A: Pharmacokinetics (PK): Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of Total Radioactivity in Plasma and Whole Blood Following a Single Oral Dose of [14C]-LY3866288 | Predose up to Day 21 postdose
Part A: PK: Maximum Observed Plasma Concentration (Cmax) of LY3866288 in Plasma Following a Single Oral Dose of [14C]-LY3866288 | Predose up to Day 7 postdose
Part A: PK: Maximum Observed Plasma Concentration (Cmax) of Total Radioactivity in Plasma and Whole Blood Following a Single Oral Dose of [14C]-LY3866288 | Predose up to Day 21 postdose
Part A: PK: Ratio of AUC0-inf of Plasma LY3866288 to AUC0-inf of Plasma Total Radioactivity | Predose up to Day 21 postdose
Part A: PK: Ratio of AUC0-inf of Whole Blood Total Radioactivity to AUC0-inf of Plasma Total Radioactivity | Predose up to Day 21 postdose
Part B: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of LY3866288 in Plasma | Predose up to Day 9 postdose
Part B: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of [14C]-LY3866288 in Plasma | Predose up to Day 9 postdose
Part B: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of Total Radioactivity in Plasma | Predose up to Day 9 postdose
Part B: PK: Maximum Observed Plasma Concentration (Cmax) of LY3866288 in Plasma | Predose up to Day 9 postdose
Part B: PK: Maximum Observed Plasma Concentration (Cmax) of [14C]-LY3866288 in Plasma | Predose up to Day 9 postdose
Part B: PK: Maximum Observed Plasma Concentration (Cmax) of Total Radioactivity in Plasma | Predose up to Day 9 postdose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No